CLINICAL TRIAL: NCT01631851
Title: Cognitive-Behavioral Therapy for Irritability in Adolescents With High Functioning Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0102012121-B
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Autism; Autism Spectrum Disorder (ASD; Asperger's Disorder; Pervasive Developmental Disorder (PDD-NOS)
Keywords: Autism; Irritability; Disruptive Behavior; Aggression; Behavior Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Asperger Syndrome; Child Development Disorders, Pervasive; Problem Behavior; Aggression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive behavior therapy (Experimental)
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT) for Irritability

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT) for Irritability — CBT is an individually administered behavioral interventions aimed at reducing irritability and disruptive behavior. There are 10 to 12 weekly sessions that are conducted with the child and the parent. During these sessions children are taught to recognize antecedents and consequences of problem behavior and to use emotion regulation and problem-solving skills to reduce irritability, aggression and noncompliance.
  Other Names: Anger Control Training

SUMMARY:
In addition to the core symptoms, children and adolescents with Autism Spectrum Disorder (ASD) often exhibit disruptive behavior problems including irritability, tantrums, noncompliance, and aggression. This is a pilot study of Cognitive-Behavioral Therapy, also known as Anger Control Training, in adolescents with high-functioning ASD. CBT teaches children to recognize antecedents and consequences of problem behavior and to use emotion regulation and problem-solving skills to reduce irritability, aggression and noncompliance. This form of CBT has been well-studied in typically developing children with disruptive behavior and we are investigating if this treatment can be feasible and helpful, with appropriate modifications, for irritability and disruptive behavior in ASD.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of autistic disorder, Asperger's disorder, or PDD-NOS
* presence of disruptive behaviors such as irritability and anger outbursts
* IQ above 80
* Unmedicated or on stable medication

Exclusion Criteria:

* medical or psychiatric condition that would require alternative treatment

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04-23 (Actual); Study Completion 2013-04-23 (Actual)

PRIMARY OUTCOMES:
ABC Irritability Scale | 1 week
  Parent rating of irritability and disruptive behavior that has been often used in studies with children with ASD

CONTACTS AND LOCATIONS:
Overall Officials: Denis Sukhodolsky, Ph.D., Principal Investigator — Yale University, Child Study Center
Locations (1):
- Yale Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Sukhodolsky DG, Vitulano LA, Carroll DH, McGuire J, Leckman JF, Scahill L. Randomized trial of anger control training for adolescents with Tourette's syndrome and disruptive behavior. J Am Acad Child Adolesc Psychiatry. 2009 Apr;48(4):413-421. doi: 10.1097/CHI.0b013e3181985050. PMID 19242384
- [Background] Aman MG, McDougle CJ, Scahill L, Handen B, Arnold LE, Johnson C, Stigler KA, Bearss K, Butter E, Swiezy NB, Sukhodolsky DD, Ramadan Y, Pozdol SL, Nikolov R, Lecavalier L, Kohn AE, Koenig K, Hollway JA, Korzekwa P, Gavaletz A, Mulick JA, Hall KL, Dziura J, Ritz L, Trollinger S, Yu S, Vitiello B, Wagner A; Research Units on Pediatric Psychopharmacology Autism Network. Medication and parent training in children with pervasive developmental disorders and serious behavior problems: results from a randomized clinical trial. J Am Acad Child Adolesc Psychiatry. 2009 Dec;48(12):1143-54. doi: 10.1097/CHI.0b013e3181bfd669. PMID 19858761